CLINICAL TRIAL: NCT02256813
Title: A Study to Evaluate the Effect of Multiple Doses of 500 mg of BIRT 2584 XX Tablets on the Pharmacokinetic Parameters of Warfarin, Omeprazole, Caffeine, and Dextromethorphan Dosed Orally and Midazolam Dosed IV, in Healthy Male Volunteers
Brief Title: Study to Evaluate the Effect of Multiple Doses of BIRT 2584 XX Tablets on the Pharmacokinetic Parameters of Warfarin, Omeprazole, Caffeine, and Dextromethorphan in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1206.10
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Warfarin; Omeprazole; Dextromethorphan; Caffeine; Midazolam; Vitamin K 1

ARMS (1):
- BIRT 2584 XX + PK-cocktail (Experimental)
  Interventions: Drug: BIRT 2584 XX; Drug: Warfarin sodium; Drug: Omeprazole; Drug: Dextromethorphan hydrobromide; Drug: Caffeine; Drug: Midazolam hydrochloride; Drug: Vitamin K1

INTERVENTIONS:
Drug: BIRT 2584 XX
Drug: Warfarin sodium
  Other Names: Coumadin®
Drug: Omeprazole
  Other Names: Omeprazole-ratiopharm® NT
Drug: Dextromethorphan hydrobromide
  Other Names: Hustenstiller-ratiopharm®
Drug: Caffeine
  Other Names: Coffeinum®
Drug: Midazolam hydrochloride
  Other Names: Dormicum®
Drug: Vitamin K1
  Other Names: Konakion®

SUMMARY:
The study aimed to investigate the effect of BIRT 2584 XX and its metabolite BI 610100 on the Pharmacokinetics (PK) of five probe substrates for cytochrome P450 isozymes.

The substrates used to monitor enzyme activity were oral warfarin (for CYP2C9), oral omeprazole (for CYP2C19), oral dextromethorphan (for CYP2D6), oral caffeine (for CYP1A2) and intravenous midazolam (for hepatic CYP3A)

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 and ≤55 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2
* healthy male subjects as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead ECG at the screening visit
* signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* non-smoker (a subject is considered to be a non-smoker if he has never smoked or has stopped smoking ≥ 6 months before the screening visit)
* agree not to take any prescription medications or non-prescription drugs (including herbal preparations and vitamins) without approval by the investigator and not to receive vaccinations during the course of the study
* agree not to eat oranges, grapefruits, broccoli, Brussels sprouts, or char grilled meats and not to drink grapefruit juice during the course of the study
* agree not to drink alcoholic beverages during the course of the study
* agree not to drink or eat caffeine and theobromine containing beverages and foods during the course of the study

Exclusion Criteria:

* any finding of the medical examination (including Blood Pressure, Pulse Rate, and ECG) deviating from normal and of clinical relevance
* gastrointestinal, hepatic, renal, respiratory (e.g. asthma), cardiovascular, metabolic, immunologic, haematological, oncological, or hormonal disorders
* any surgical or medical condition that could interfere with the administration of the study drug or interpretation of the study results
* diseases of the Central nervous system (CNS) (such as epilepsy) or psychiatric disorders or neurological disorders
* relevant history of orthostatic hypotension, fainting spells, or blackouts
* chronic or relevant acute infections
* history of allergy/hypersensitivity (including drug allergy) considered relevant to the trial as judged by the investigator
* immunisation during the 2 weeks prior to the screening visit
* known intolerance to benzodiazepines
* known intolerance to the active and/or inactive ingredients in caffeine, warfarin, vitamin K1, omeprazole, or dextromethorphan
* known acute angle-closure glaucoma
* elevated prothrombin time as determined by Prothrombin time (INR) > 1.3
* intake of drugs with a long half-life (greater than 24 hrs) (less than one month prior to administration or during the trial)
* use of any drugs which might influence the results of the trial (less than 10 days prior to study drug administration or expected during the trial)
* use of chewing tobacco or nicotine replacement devices within 6 months before the screening visit
* participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* alcohol abuse (more than 60 g of ethanol per day)
* blood donation or loss greater than 100 mL (less than one month prior to administration or expected during the trial)
* clinically relevant laboratory abnormalities

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
AUC0-inf (Area under the concentration-time curve of midazolam IV and S-warfarin in plasma over the time interval from 0 extrapolated to infinity) | up to day 19
AUC (Area under the concentration-time curve of the ratio of omeprazole to 5-hydroxyomeprazole in plasma) | up to day 19
0-12 hr urinary molar ratio of caffeine metabolites (1-Methylxanthine + 1-Methylurate +5-Acetylamino-6-formylamino-3-methyluracil)/ 1,7-Dimethylurate | up to 12 hours after administration
0-12 hr urinary dextromethorphan/dextrorphan ratio | up to 12 hours after administration

SECONDARY OUTCOMES:
AUC0-tz (Area under the concentration-time curve of the S-warfarin, omeprazole and midazolam IV in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to day 19
Cmax (Maximum measured concentration of the S-warfarin, omeprazole and midazolam IV in plasma) | up to day 19
tmax (Time from dosing to the maximum concentration of the S-warfarin, omeprazole and midazolam IV in plasma) | up to day 19
λz (Terminal rate constant of the S-warfarin, omeprazole and midazolam IV in plasma) | up to day 19
t1/2 (Terminal rate constant of the S-warfarin, omeprazole and midazolam IV in plasma) | up to day 19
MRT (Mean residence time of the S-warfarin, omeprazole and midazolam IV in the body after administration) | up to day 19
CL/F (Apparent clearance of the S-warfarin, omeprazole and midazolam IV in plasma after extravascular single dose administration) | up to day 19
Vz/F (Apparent volume of distribution during the terminal phase λz following extravascular administration S-warfarin, omeprazole and midazolam IV) | up to day 19
AUC0-inf (Area under the concentration-time curve of omeprazole in plasma over the time interval from 0 extrapolated to infinity) | up to day 19
trough levels of BIRT 2584 XX and BI 610100 | up to day 19
approximate peak levels of BIRT 2584 XX and BI 610100 | up to day 19
Number of subjects with adverse events | up to 48 days
Number of subjects with abnormal changes in laboratory parameters | up to 48 days